CLINICAL TRIAL: NCT03967860
Title: Role of Post Surgery CT Following Laparoscopic Vertical Sleeve Gastrectomy
Acronym: LSG-CT
Status: Completed | Type: Observational
Sponsor: Francesco De Cobelli (Other)
Responsible Party: Sponsor-Investigator, Francesco De Cobelli, Professor of Radiology, Director of Specialiaztion School in Radiology, Head of Clinical and Experimental Radiology, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: LSG-CT
Record Dates: First submitted 2019-04-02; First posted 2019-05-30 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Obesity
Keywords: CT Scan
MeSH Terms: conditions — Obesity | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CT scan — Post surgical standard CT Scan as predictor of complication

SUMMARY:
Obesity is a extremely widespread condition in Europe and North America, burdened by a series of complications characterized by major morbidity and morbility. In recent years, bariatric surgery has progressively assumed a leading role in the treatment of morbid obesity and restrictive bariatric surgery procedures, such as laparoscopic vertical sleeve gastrectomy are common.

The aim of the study is to retrospectively determine the value of postoperative CT after LSG as an early tool to identify risk factors for the subsequent development of gastric fistula and enable to stratify postoperative risk in asymptomatic patients and ensure effective management of these risk factors.

ELIGIBILITY:
Inclusion Criteria:

* adult obese patients with LSG
* BMI ≥ 40 kg/m2 or BMI between 35 and 40 kg/m2
* evidence of obesity related comorbidity
* availability of upper abdomen CT scan with IV and oral contrast medium within 72 hours of surgery

Exclusion Criteria:

* Pregnant women
* allergy to contract medium
* lack of venous access
* patients who did not have a post-surgical upper abdomen CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients with BMI ≥ 40 kg/m2 or between 35 e 40 kg/m2 with evidence of obesity related comorbidity
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
Value of Post surgery CT in identifying risks for subsequent development of gastric fistula | 72 hours post LSG
  Measurements of: presence or abscence of fistula and site; presence/abscence of hematoma and site; presence/abscence of gastric torsion; Stapler to pylorus distance and stapler length

SECONDARY OUTCOMES:
Post surgery risk | 72 hours post LSG
  Risk stratification based on the correlation of the measurements obtained from the primary objective on outcome (complication vs non complication).

CONTACTS AND LOCATIONS:
Locations (1):
- Deaprtment of Radiology, IRCCS Ospadale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No